CLINICAL TRIAL: NCT02723123
Title: Respiratory Behaviour of Extremely Preterm Infants Receiving Non-invasive Respiratory Support During the Immediate Post-extubation Period
Brief Title: Non-invasive Support in Extremely Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guilherme Sant'Anna, MD (Other)
Responsible Party: Sponsor-Investigator, Guilherme Sant'Anna, MD, Assistant Professor, Department of Paediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NIVNAVA 01
Record Dates: First submitted 2015-11-27; First posted 2016-03-30 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Noninvasive Ventilation
Keywords: CPAP; NIPPV; Extubation failure; Cardiorespiratory behaviour; NIV-NAVA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPAP (Experimental): CPAP will be provided for a approximately 45 minutes.
  Interventions: Other: Recording of cardio-respiratory signals
- NIPPV (Experimental): NIPPV will be provided for a approximately 45 minutes.
  Interventions: Other: Recording of cardio-respiratory signals
- NIV-NAVA (Experimental): NIV-NAVA will be provided for a approximately 45 minutes.
  Interventions: Other: Recording of cardio-respiratory signals

INTERVENTIONS:
Other: Recording of cardio-respiratory signals — Biological signals: ECG, RIP, SpO2 and Pulse rate will be recorded during the interventions and analyzed offline.

SUMMARY:
Non-invasive respiratory support is routinely provided to extremely preterm infants following disconnection from mechanical ventilation, in the form of continuous positive airway pressure (CPAP) or non-invasive positive pressure ventilation (NIPPV). However, these modes remain sub-optimal due to lack of synchronization and upper airway defensive mechanisms that potentially hinder their effectiveness. Non-invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA) is a novel mode that may overcome some of these problems but has not been investigated in this population. Investigators hypothesize that there will be significant differences in cardiorespiratory behavior in extremely preterm infants receiving CPAP, NIPPV and NIV-NAVA during the immediate post-extubation period.

DETAILED DESCRIPTION:
A large proportion of extremely preterm infants are mechanically ventilated through the use of endotracheal intubation. However, clinicians try to avoid intubation due to the complications that may arise from being mechanically ventilated such as ventilator associated pneumonia (VAP), pulmonary hemorrhage, air leak etc. In order to the prevent these complications, clinicians accelerate weaning and provide non-invasive respiratory support. The most commonly used type of non-invasive respiratory support following extubation is nasal continuous positive airway pressure (NCPAP). NCPAP has been shown to improve oxygenation, reduce airway resistance, increase tidal volume, stabilize chest wall and maintain functional residual capacity. In addition to NCPAP, nasal intermittent positive pressure ventilation (NIPPV) has become a popular choice as a post-extubation respiratory support mode. However, there is a lack of knowledge regarding the effects of synchronization between the infant's own spontaneous respiratory efforts and ventilator inflations.

Synchronization, especially during non-invasive ventilation, is difficult to achieve in preterm infants due to their rapid respiratory rates, short inspiratory times, periodic breathing, leaks and small tidal volumes. Previous studies have used devices such as an abdominal capsule to allow for synchronization while the infant is receiving NIPPV. The abdominal capsule itself is prone to incorrect placement, time delays and ineffective synchronization. Neurally Activated Ventilatory Assistance (NAVA) is a new technology that can be used during invasive and non-invasive ventilation. In this novel mode, the electrical activity of the diaphragm, called EAdi, is detected be electrodes inserted at the tip of a specialized nasogastric tube. The EAdi represents the patient's inherent neural respiratory drive. The ventilator assists each spontaneous breath by delivering pressure that is linearly proportional to the EAdi. The mechanical breath is initiated at the start of diaphragmatic contraction and maintained until the EAdi is at 60 to 70% of the peak pressure generated. Therefore, the inspiratory time, expiratory time and peak inflation pressure are all controlled and determined by the patient, providing patient-ventilator synchrony.

ELIGIBILITY:
Inclusion Criteria:

* birth weight under 1250 grams receiving invasive mechanical ventilation

Exclusion Criteria:

* infants with major congenital anomalies, congenital heart defects, neuromuscular disease, diaphragmatic paralysis or palsy, diagnosed phrenic nerve injury, esophageal perforation, hemodynamic instability as well as infants on interpose, narcotics or sedative agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Differences on cardiorespiratory behaviour in extremely preterm infants receiving CPAP, NIPPV and NIV-NAVA | Immediate post-extubation period (30 minutes after extubation)
  Cardiorespiratory signals (ECG, thoraco-abdominal movements, oxygen saturation and TcPCO2), and ventilator signals (pressure and EAdi waveforms, tidal volume, MAP, PIP, PEEP, and FiO2) will continuously be measured throughout the recordings. Analysis of these signals will be performed offline. From these cardiorespiratory signals, behaviour will be analyzed by calculations of: cardiorespiratory variability, respiratory pauses, thoraco-abdominal asynchrony, respiratory movement artifacts and regular breathing pattern.
  Cardiorespiratory behavior will be calculated using the instantaneous power estimate of all respiratory and cardiac signals computed. To this end, each of the continuous metrics will be squared and averaged over a symmetric, two-sided window of length. For example, the correlation between respiratory and heart rates will be estimated by averaging the product fmax*hmax over the same window.

SECONDARY OUTCOMES:
Differences on in patient-ventilator interaction in extremely preterm infants receiving CPAP, NIPPV and NIV-NAVA | Immediate post-extubation period (30 minutes after extubation)
  Patient-ventilator interaction which will be analyzed by calculating the following parameters: Trigger delay, cycling off delay, number of breaths with premature cycling off, asynchrony index, wasted inspiratory efforts, relationship and proportionality between ventilator assist and patient respiratory demand.
  Despite the different units of measure for the aforementioned parameters, these values together will represent an accurate description of the interaction between the patient and the ventilator. These parameters will compared between the three modes.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Sant'Anna, MD, Study Chair — McGill University; Wissam Shalish, MD, Principal Investigator — McGill University; Robert Kearney, PhD, Principal Investigator — McGill University; Karen Brown, MD, Principal Investigator — McGill University; Doina Precup, PhD, Principal Investigator — McGill University
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada